CLINICAL TRIAL: NCT04696549
Title: Art Museum Program for Seniors With Cognitive Disorders and Care-partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00267702
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Dementia
Keywords: dementia; caregiving; self-esteem
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual visual art experience for individuals with dementia and their family care-partners (Experimental): Individuals with dementia and their family care-partners will participate in three monthly one-hour virtual art sessions in which the facilitator uses Visual Thinking Strategies technique to facilitate participants' viewing and discussion about virtual art images.
  Interventions: Behavioral: Virtual visual art experience guided by Visual Thinking Strategies

INTERVENTIONS:
Behavioral: Virtual visual art experience guided by Visual Thinking Strategies — All study dyads (where study dyad consists of a participant with dementia and his/her care-partner) will participate in 3 scheduled virtual visual art sessions via Zoom. Each session will last about an hour and will include a guided discussion of pre-selected visual art using the Visual Thinking Strategies approach. It is anticipated that two pieces of art will be shown during each art session. The three sessions will be scheduled one month apart.

SUMMARY:
As the population ages, there is increasing interest in developing innovative approaches to promote and sustain mental and emotional well-being. Recent studies have linked engagement with the arts with supporting cognitive functioning, promoting empathy and greater sense of life purpose. The need to develop alternative approaches to sustain emotional well-being is especially acute for the nearly 6 million older Americans who suffer from Alzheimer's disease. There is a need for quality activities that can be done virtually for homebound individuals with cognitive disorders and the individuals' family care-partners.

The investigators intend to institute a 3-session virtual art museum pilot program for seniors with cognitive disorders and care-partners using the Visual Thinking Strategies approach. The investigators hypothesize that participation in a virtual guided visual arts experience will enhance emotional well-being and self-esteem for both seniors with cognitive impairment and the seniors' care-partners.

DETAILED DESCRIPTION:
A number of innovative programs currently exist nationally that are exploring ways to connect to connect older adults with cognitive impairment with the arts. One example is the "Meet Me at MOMA" program at the Museum of Modern Art (MOMA) in New York City, which ran a monthly program for adults with dementia and the adults' care-partners. Researchers studying this program found that participants benefited in terms of improvement in measures of well-being, including higher ratings on scales looking at self-esteem and quality of life . Additionally, other art-based interventions have shown improvements in well-being and mood for the care-partners of individuals with dementia.

One well-validated approach to engaging individuals with works of visual art is "Visual Thinking Strategies". Visual Thinking Strategies (VTS) uses a structured technique to guide viewers to engage with visual art that builds on lived experiences and does not presuppose any knowledge of art or art history. Previous work has utilized Visual Thinking Strategies in educational settings and for clinicians to promote professional identity formation. It has not been studied in clinical settings with patients or with individuals with cognitive disorders. Yet, this approach may have particular benefits for elders with cognitive impairment as it encourages the elders' engagement in the "here and now" and therefore, also provides immediate positive feedback and validation to participants. As such, Visual Thinking Strategies has the potential to contribute to emotional well-being, self-esteem, and meaning for older adults with cognitive impairment.

Subjects: The Johns Hopkins Club Memory Group consists of about 25 older adults with cognitive disorders and the older adults' family care-partners. This group meets twice monthly for social interaction and engagement and is led by senior nurse, Andrea Nelson, Registered Nurse (RN). As this will be a small pilot program, individuals with cognitive disorders and the individuals' care-partners will be individually invited to participate in the program by Andrea Nelson, RN. The investigators intend to recruit a total of 4-6 individuals with early to moderate cognitive impairment and the individuals' care-partners for this pilot program.

Consent process:

Andrea Nelson, Registered Nurse, will obtain telephone consent from both the individuals with cognitive disorder and the individuals' family care-partners. For those individuals who agree to participate, Andrea Nelson, Registered Nurse will screen for eligibility and will do a Clinical Dementia Rating Scale determination by telephone. Participants will receive a written copy of the study by mail.

Study plan:

All study dyads will participate in 3 scheduled Visual Thinking Strategies sessions via Zoom. Each session will last about an hour and will include a guided discussion of pre-selected visual art using the Visual Thinking Strategies approach. It is anticipated that two pieces of art will be shown during each session. The three sessions will be scheduled one month apart. In advance of each session, participants will be mailed the study instruments listed below along with an addressed, stamped envelope to mail the completed forms back to Andrea Nelson, Registered Nurse upon completion.

Immediately prior to the start of each Visual Thinking Strategies art session, both members of the study dyad will be asked to complete the following scales.

1. Rosenberg Self-Esteem Scale- This is a 10-item self-report scale with items answered on a 4-point Likert scale from strongly agree to strongly disagree. Although originally developed for adolescents, it is considered to be a valid tool for self-esteem assessment in adults.
2. Smiley Face Mood Rating Scale- A pictorial self-report Likert scale with 5 smiley faces ranging from very unhappy to very happy Immediately following each art session, both members of the study dyad will be asked to complete another Smiley Face Mood Rating Scale.

In addition, after each art session, a feedback questionnaire will be completed by the individual with cognitive disorder and a separate feedback questionnaire will be completed by the care-partner. The feedback questionnaires will be completed anytime in the subsequent 2 days following the VTS session. The questionnaires solicit feedback about how enjoyable the art session was and what changes in emotional well-being were experienced as a result of the art session participation.

Participants will return the completed Rosenberg Self-Esteem Scales, Smiley Face Mood Rating Scales, and post-session questionnaires in an addressed, stamped envelope to Andrea Nelson, Registered Nurse.

ELIGIBILITY:
Inclusion Criteria:

* Club Memory member with cognitive disorder and family care-partner. This will constitute a study dyad.
* Early to moderate cognitive impairment, as evidenced by Clinical Dementia Rating scale of 0.5-2.0. The Clinical Dementia Rating scale is a clinical rating scale used for dementia staging based on 6 domains of functioning that will be performed by Andrea Nelson, Registered Nurse, and is part of normal dementia care in the Johns Hopkins Bayview Memory and Alzheimer's Treatment Center. A rating of 0=normal, 0.5= mild cognitive impairment, 1.0=mild dementia, 2.0=moderate dementia, 3.0=severe dementia.
* Care-partner access to laptop or iPad and comfort with using Zoom technology
* Agreement by individual with cognitive disorder and care-partner to participate in all 3 Visual Thinking visual art sessions
* Agreement by individual with cognitive disorder and care-partner to participate in the study and complete questionnaires before and after each session

Exclusion Criteria:

* Non-English speaker
* Clinical Dementia Rating higher than 2.0 for individual with cognitive impairment
* Inability to use a laptop or iPad for Zoom sessions

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Change in self-esteem as assessed by the Rosenberg Self-Esteem Scale | At first session and third session, up to 3 months
  Impact of participation in a virtual art museum program on both older adults with cognitive disorders and their care-partners on survey measure of self-esteem. The Rosenberg Self-Esteem Scale is a 10-item self-report scale. Each item response is scored on a 4-point Likert Scale where 1 = Strongly agree and 4= Strongly disagree. Higher scores indicate higher self-esteem, and lower scores indicate lower self-esteem.
Change in self-report mood as assessed by the Smiley Face Mood Rating Scale | Before and immediately after each visual art session, up to 3 months
  Impact of participation in a virtual art museum program on both older adults with cognitive disorders and their care-partners on self-report measure of mood. Smiley Face Mood Rating Scale- A pictorial self-report Likert scale with 5 smiley faces ranging from very unhappy (scored as 1), to very happy (scored as 5). Higher scores indicate a more positive mood and lower scores indicate a more negative mood.

SECONDARY OUTCOMES:
to get feedback from family care-partners about their experience in participating in a virtual art museum program regarding satisfaction with a virtual program of this nature | up to 48 hours after first visual art session
  Post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 7 question items, 3 of which are YES/NO response, 2 of which are multiple choice response, one is a 10-point rating scale for satisfaction level where 10 is "very high satisfaction" and 1 is "very low satisfaction". One question is open-narrative free response.
to get feedback from family care-partners about their experience in participating in a virtual art museum program regarding acceptability and satisfaction with a virtual program of this nature | up to 48 hours after second visual art session
  post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 7 question items, 3 of which are YES/NO response, 2 of which are multiple choice response, 1 is a 10-point rating scale for satisfaction level where is "very high satisfaction" and 1 is "very low satisfaction". One question is open-narrative free response
to get feedback from family care-partners about their experience in participating in a virtual art museum program regarding acceptability and satisfaction with a virtual program of this nature | up to 48 hours after third visual art session
  post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 7 question items, 3 of which are YES/NO response, 2 of which are multiple choice response, 1 is a 10-point rating scale for satisfaction level where is "very high satisfaction" and 1 is "very low satisfaction". One question is open-narrative free response
to get feedback from individuals with cognitive disorders about their experience in participating in a virtual art museum program regarding acceptability and satisfaction with a virtual program of this nature | up to 48 hours after first visual art session
  post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 6 question items. 5 items are YES/NO response, and 1 item is multiple choice response
to get feedback from individuals with cognitive disorders about their experience in participating in a virtual art museum program regarding acceptability and satisfaction with a virtual program of this nature | up to 48 hours after second visual art session
  post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 6 question items. 5 items are YES/NO response, and 1 item is multiple choice response
to get feedback from individuals with cognitive disorders about their experience in participating in a virtual art museum program regarding acceptability and satisfaction with a virtual program of this nature | up to 48 hours after third visual art session
  post-visual art experience questionnaire asking questions about satisfaction. The questionnaire consists of 6 question items. 5 items are YES/NO response, and 1 item is multiple choice response

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Lehmann, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No